CLINICAL TRIAL: NCT01931670
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Elagolix in Subjects With Moderate to Severe Endometriosis-Associated Pain
Brief Title: A Global Phase 3 Study to Evaluate the Safety and Efficacy of Elagolix in Subjects With Moderate to Severe Endometriosis-Associated Pain
Acronym: ELARIS EM-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-671; 2011-004295-11 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-03

CONDITIONS: Endometriosis
Keywords: Non-Menstrual Pelvic Pain (NMPP); Dysmenorrhea (DYS); Elagolix; Endometriosis Associated Pain; Gonadotropin-Releasing Hormone Antagonist
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo twice daily (BID) for the 6-month Treatment Period
  Interventions: Other: placebo
- Elagolix 150 mg QD (Experimental): Elagolix 150 mg once daily (QD) for the 6-month Treatment Period
  Interventions: Drug: Elagolix
- Elagolix 200 mg BID (Experimental): Elagolix 200 mg BID for the 6-month Treatment Period
  Interventions: Drug: Elagolix

INTERVENTIONS:
Other: placebo
  Arms: Placebo
Drug: Elagolix
  Other Names: ABT-620; elagolix sodium
  Arms: Elagolix 150 mg QD; Elagolix 200 mg BID

SUMMARY:
A randomized study evaluating the safety and efficacy of elagolix in the management of moderate to severe endometriosis-associated pain in adult premenopausal female subjects.

DETAILED DESCRIPTION:
The study consists of 4 periods: 1) Washout Period (if applicable); 2) a Screening Period of up to 100 days prior to first dose; 3) a 6 month Treatment Period; and 4) a Post treatment Follow-up Period of up to 12 months (if applicable). An electronic diary will be dispensed and training provided to record endometriosis-associated pain, uterine bleeding, and analgesic medication use for endometriosis-associated pain on a daily basis. Pregnancy testing will be performed monthly throughout the study. Subjects will be required to use nonhormonal dual contraception during the study, and will be counseled on appropriate and effective forms of birth control to promote pregnancy prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal female, between 18 and 49 years of age, inclusive, at the time of signing consent.
2. Clinical diagnosis of endometriosis (laparoscopy or laparotomy) performed within 10 years of entry into the Washout Period.
3. Agrees to use required birth control methods during the entire length of participation in the study.
4. Subject has a Composite Pelvic Signs and Symptoms Score total score of 6 or greater at Screening with a score of at least 2 for dysmenorrhea AND at least 2 for non-menstrual pelvic pain.
5. Subjects must have at least two regular menstrual cycles with an interval of 24-38 days within the Screening Period, prior to Day 1.

Exclusion Criteria:

1. Subject is pregnant or breast feeding or is planning a pregnancy within the next 24 months or is less than 6 months postpartum, post-abortion, or post-pregnancy at the time of entry into the Screening Period.
2. Subject has a history of previous non-response to gonadotropin-releasing hormone (GnRH) agonists, GnRH antagonists, Depot medroxyprogesterone acetate, or aromatase inhibitors as assessed by subject report of no improvement in dysmenorrhea or non-menstrual pelvic pain.
3. Subject has chronic pelvic pain that is not caused by endometriosis that requires chronic analgesic or other chronic therapy, or that would interfere with the assessment of endometriosis related pain.
4. Clinically significant gynecologic condition identified on Screening transvaginal ultrasound or endometrial biopsy.
5. Subject has a history of osteoporosis or other metabolic bone disease.
6. Subject has a current history of undiagnosed abnormal uterine bleeding.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 815 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taylor HS, Giudice LC, Lessey BA, Abrao MS, Kotarski J, Archer DF, Diamond MP, Surrey E, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Rowan JP, Duan WR, Ng J, Schwefel B, Thomas JW, Jain RI, Chwalisz K. Treatment of Endometriosis-Associated Pain with Elagolix, an Oral GnRH Antagonist. N Engl J Med. 2017 Jul 6;377(1):28-40. doi: 10.1056/NEJMoa1700089. Epub 2017 May 19. PMID 28525302
- [Derived] Beck D, Winzenborg I, Liu M, Degner J, Mostafa NM, Noertersheuser P, Shebley M. Population Pharmacokinetics of Elagolix in Combination with Low-Dose Estradiol/Norethindrone Acetate in Women with Uterine Fibroids. Clin Pharmacokinet. 2022 Apr;61(4):577-587. doi: 10.1007/s40262-021-01096-w. Epub 2021 Dec 8. PMID 34878624
- [Derived] Abrao MS, Surrey E, Gordon K, Snabes MC, Wang H, Ijacu H, Taylor HS. Reductions in endometriosis-associated pain among women treated with elagolix are consistent across a range of baseline characteristics reflective of real-world patients. BMC Womens Health. 2021 Jun 16;21(1):246. doi: 10.1186/s12905-021-01385-3. PMID 34134684
- [Derived] Stodtmann S, Nader A, Polepally AR, Suleiman AA, Winzenborg I, Noertersheuser P, Ng J, Mostafa NM, Shebley M. Validation of a quantitative systems pharmacology model of calcium homeostasis using elagolix Phase 3 clinical trial data in women with endometriosis. Clin Transl Sci. 2021 Jul;14(4):1611-1619. doi: 10.1111/cts.13040. Epub 2021 May 7. PMID 33963686
- [Derived] Beck D, Winzenborg I, Gao W, Mostafa NM, Noertersheuser P, Chiuve SE, Owens C, Shebley M. Integrating real-world data and modeling to project changes in femoral neck bone mineral density and fracture risk in premenopausal women. Clin Transl Sci. 2021 Jul;14(4):1452-1463. doi: 10.1111/cts.13006. Epub 2021 Apr 8. PMID 33650259
- [Derived] Agarwal SK, Singh SS, Archer DF, Mai Y, Chwalisz K, Gordon K, Surrey E. Endometriosis-Related Pain Reduction During Bleeding and Nonbleeding Days in Women Treated with Elagolix. J Pain Res. 2021 Feb 2;14:263-271. doi: 10.2147/JPR.S284703. eCollection 2021. PMID 33564263
- [Derived] Pokrzywinski RM, Soliman AM, Snabes MC, Chen J, Taylor HS, Coyne KS. Responsiveness and thresholds for clinically meaningful changes in worst pain numerical rating scale for dysmenorrhea and nonmenstrual pelvic pain in women with moderate to severe endometriosis. Fertil Steril. 2021 Feb;115(2):423-430. doi: 10.1016/j.fertnstert.2020.07.013. Epub 2020 Oct 14. PMID 33066973
- [Derived] Abbas Suleiman A, Nader A, Winzenborg I, Beck D, Polepally AR, Ng J, Noertersheuser P, Mostafa NM. Exposure-Safety Analyses Identify Predictors of Change in Bone Mineral Density and Support Elagolix Labeling for Endometriosis-Associated Pain. CPT Pharmacometrics Syst Pharmacol. 2020 Nov;9(11):639-648. doi: 10.1002/psp4.12560. Epub 2020 Oct 8. PMID 32945631
- [Derived] Taylor HS, Soliman AM, Johns B, Pokrzywinski RM, Snabes M, Coyne KS. Health-Related Quality of Life Improvements in Patients With Endometriosis Treated With Elagolix. Obstet Gynecol. 2020 Sep;136(3):501-509. doi: 10.1097/AOG.0000000000003917. PMID 32769633
- [Derived] Winzenborg I, Polepally AR, Nader A, Mostafa NM, Noertersheuser P, Ng J. Effect of Elagolix Exposure on Clinical Efficacy End Points in Phase III Trials in Women With Endometriosis-Associated Pain: An Application of Markov Model. CPT Pharmacometrics Syst Pharmacol. 2020 Aug;9(8):466-475. doi: 10.1002/psp4.12545. Epub 2020 Jul 31. PMID 32621325
- [Derived] Surrey ES, Soliman AM, Palac HL, Agarwal SK. Impact of Elagolix on Workplace and Household Productivity Among Women with Moderate to Severe Pain Associated with Endometriosis: A Pooled Analysis of Two Phase III Trials. Patient. 2019 Dec;12(6):651-660. doi: 10.1007/s40271-019-00394-7. PMID 31654294
- [Derived] Pokrzywinski RM, Soliman AM, Chen J, Snabes M, Diamond MP, Surrey E, Coyne KS. Impact of elagolix on work loss due to endometriosis-associated pain: estimates based on the results of two phase III clinical trials. Fertil Steril. 2019 Sep;112(3):545-551. doi: 10.1016/j.fertnstert.2019.04.031. Epub 2019 Jun 18. PMID 31227284
- [Derived] Rolla E. Endometriosis: advances and controversies in classification, pathogenesis, diagnosis, and treatment. F1000Res. 2019 Apr 23;8:F1000 Faculty Rev-529. doi: 10.12688/f1000research.14817.1. eCollection 2019. PMID 31069056
- [Derived] Wang ST, Johnson SJ, Mitchell D, Soliman AM, Vora JB, Agarwal SK. Cost-effectiveness of elagolix versus leuprolide acetate for treating moderate-to-severe endometriosis pain in the USA. J Comp Eff Res. 2019 Apr;8(5):337-355. doi: 10.2217/cer-2018-0124. Epub 2019 Feb 6. PMID 30724096
- [Derived] Winzenborg I, Nader A, Polepally AR, Liu M, Degner J, Klein CE, Mostafa NM, Noertersheuser P, Ng J. Population Pharmacokinetics of Elagolix in Healthy Women and Women with Endometriosis. Clin Pharmacokinet. 2018 Oct;57(10):1295-1306. doi: 10.1007/s40262-018-0629-6. PMID 29476499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 187 sites in Argentina, Austria, Australia, Brazil, Czech Republic, Hungary, Italy, New Zealand, Poland, South Africa, Spain, the United States, and the United Kingdom.
Pre-assignment Details: The study consisted of 4 periods: a Washout Period (if applicable); a Screening Period of ≤ 100 days prior to first dose; a 6-month Treatment Period; and a Post-Treatment Follow-up Period of ≤ 12 months (if applicable). Participants were randomized into the study in a 3:2:2 ratio to placebo, elagolix 150 mg QD, or elagolix 200 mg BID, respectively.
Period: Treatment Period
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Started | 360 | 226 | 229
Completed | 270 | 178 | 184
Not Completed | 90 | 48 | 45
Not completed — Exclusionary Medication Received | 1 | 1 | 1
Not completed — Surgery/Invasive Intervention | 4 | 2 | 0
Not completed — Subject Noncompliant | 4 | 9 | 5
Not completed — Adverse Event | 19 | 8 | 21
Not completed — Lack of Efficacy | 11 | 2 | 2
Not completed — Pregnancy | 7 | 2 | 0
Not completed — Other | 8 | 7 | 2
Not completed — Consent Withdrawn by Subject | 17 | 12 | 7
Not completed — Lost to Follow-up | 19 | 5 | 7
Period: Post-Treatment Follow-Up (PTFU) Period
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Started (Participants who elected to enter the PTFU Period in this study for up to an additional 12 months.) | 61 | 40 | 54
Completed PTFU Month 6 | 42 | 24 | 18
Completed PTFU Month 12 | 0 | 4 | 15
Completed | 42 | 28 | 33
Not Completed | 19 | 12 | 21
Not completed — Exclusionary Medication Received | 3 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Surgery/Invasive Intervention | 4 | 4 | 2
Not completed — Other | 6 | 3 | 3
Not completed — Consent Withdrawn by Subject | 6 | 3 | 13
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo BID for the 6-month Treatment Period
- Elagolix 150 mg QD: Elagolix 150 mg QD for the 6-month Treatment Period
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID | Total
Number analyzed (Participants) | 360 | 226 | 229 | 815
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (6.69) | 33.1 (6.80) | 33.4 (6.67) | 33.2 (6.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 226 | 229 | 815
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at Month 3 Based on Daily Assessment of Dysmenorrhea (DYS)
Description: The DYS pain scale ranges from 0 (none) to 3 (severe) as recorded in a daily electronic diary. The criteria for defining a participant as a responder included a reduction of -0.85 or greater from Baseline in DYS pain as well as no increased rescue analgesic use for endometriosis-associated pain.
Time Frame: At Month 3 of the Treatment Period
Population: The modified intent-to-treat (mITT) analysis set; all randomized participants who took at least 1 dose of randomized, double-blind study drug. Population included mITT participants who either had data during the Month 3 35-day window or who prematurely discontinued prior to or at Month 3 and met the rules for last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 353 | 221 | 225
percentage of participants | 22.7 | 43.4 | 72.4
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic — An elagolix dose group was to be considered more efficacious than placebo for the co-primary endpoints if and only if both co-primary endpoints (DYS and NMPP) were statistically significant for the elagolix dose group at the 0.025 significance level
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Responders at Month 3 Based on Daily Assessment of Non-Menstrual Pelvic Pain (NMPP)
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe) as recorded in a daily electronic diary. The criteria for defining a participant as a responder included a reduction of -0.43 or greater from Baseline in NMPP as well as no increased rescue analgesic use for endometriosis-associated pain.
Time Frame: At Month 3 of Treatment Period
Population: The mITT analysis set; all randomized participants who took at least 1 dose of randomized, double-blind study drug. Population included mITT participants who either had data during the Month 3 35-day window or who prematurely discontinued prior to or at Month 3 and met the rules for last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 353 | 221 | 225
percentage of participants | 36.5 | 49.8 | 57.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.003, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline to Month 3 in Numeric Rating Scale (NRS) Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 3 of the Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 312 | 204 | 209
units on a scale | -1.33 (0.097) | -1.90 (0.122) | -2.55 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 1 of 7; Test type: Superiority; p < 0.001, mixed-effects model — For an elagolix dose group to be considered statistically significantly better than placebo on a secondary endpoint, the P value must have been ≤ 0.025 for that endpoint, for all higher-ranking secondary endpoints, and for the co-primary endpoints; Difference in LS Mean Change = -0.57, Standard Error of Mean 0.156
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 1 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -1.22, Standard Error of Mean 0.156

4. Secondary Outcome: Change From Baseline to Month 6 in DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 273 | 185 | 187
units on a scale | -0.52 (0.047) | -1.06 (0.057) | -1.65 (0.057)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 2 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.54, Standard Error of Mean 0.074
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 2 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -1.13, Standard Error of Mean 0.074

5. Secondary Outcome: Change From Baseline to Month 6 in NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 273 | 185 | 187
units on a scale | -0.48 (0.035) | -0.63 (0.044) | -0.80 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 3 of 7; Test type: Superiority; p = 0.009, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.15, Standard Error of Mean 0.056
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 3 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.32, Standard Error of Mean 0.056

6. Secondary Outcome: Change From Baseline to Month 3 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: Permitted rescue medications included the nonsteroidal anti-inflammatory drug naproxen (500 or 550 mg), and one country-specific narcotic analgesic (5 mg hydrocodone + 300 or 325 mg acetaminophen, or 30 mg codeine + 500 mg acetaminophen, or 30 mg codeine, or 37.5 mg tramadol + 325 mg acetaminophen). Assessment was based on average pill counts.
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 312 | 204 | 209
number of pills | -0.31 (0.028) | -0.36 (0.035) | -0.49 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 4 of 7; Test type: Superiority; p = 0.26, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.05, Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 4 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.18, Standard Error of Mean 0.044

7. Secondary Outcome: Change From Baseline to Month 6 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: as for outcome 6
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 273 | 185 | 187
number of pills | -0.32 (0.030) | -0.40 (0.038) | -0.52 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 5 of 7; Test type: Superiority; p = 0.088, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.08, Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 5 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.21, Standard Error of Mean 0.048

8. Secondary Outcome: Change From Baseline to Month 3 in Dyspareunia (DYSP)
Description: The DYSP pain scale ranges from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 3 of Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases. Participants who responded "not applicable" for the entire time point and at Baseline are excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 226 | 145 | 150
units on a scale | -0.30 (0.042) | -0.39 (0.052) | -0.60 (0.052)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 6 of 7; Test type: Superiority; p = 0.172, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.09, Standard Error of Mean 0.067
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 6 of 7; Test type: Superiority; p < 0.001, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.30, Standard Error of Mean 0.067

9. Secondary Outcome: Change From Baseline to Month 3 in Use of Narcotic Class of Medication (Opioids)
Description: Permitted country-specific rescue narcotic analgesics included 5 mg hydrocodone + 300 or 325 mg acetaminophen, or 30 mg codeine + 500 mg acetaminophen, or 30 mg codeine, or 37.5 mg tramadol + 325 mg acetaminophen. Assessment was based on average pill counts.
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 312 | 204 | 209
number of pills | -0.12 (0.019) | -0.12 (0.024) | -0.21 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 7 of 7; Test type: Superiority; p = 0.968, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = 0.00, Standard Error of Mean 0.030
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 7 of 7; Test type: Superiority; p = 0.007, mixed-effects model — [p-value comment as in outcome 3, analysis 1]; Difference in LS Mean Change = -0.08, Standard Error of Mean 0.030

10. Secondary Outcome: Percentage of Responders for Each Month, Except Month 3, in DYS
Description: as for outcome 1
Time Frame: Months 1, 2, 4, 5, 6 of the Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Last observation carried forward. Participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
percentage of participants
  Month 1 | 17.3 | 33.0 | 46.2
  Month 2 | 19.0 | 39.4 | 69.8
  Month 4: number analyzed (Participants) | 354 | 220 | 223
  Month 4 | 21.2 | 45.9 | 79.8
  Month 5: number analyzed (Participants) | 354 | 220 | 223
  Month 5 | 23.7 | 44.1 | 80.7
  Month 6: number analyzed (Participants) | 355 | 221 | 225
  Month 6 | 25.4 | 46.2 | 76.9
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.361, 97.5% CI 2-sided [1.507 to 3.697]
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.185, 97.5% CI 2-sided [2.707 to 6.469]
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.795, 97.5% CI 2-sided [1.811 to 4.312]
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.378, 97.5% CI 2-sided [6.615 to 16.282]
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.178, 97.5% CI 2-sided [2.084 to 4.845]
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.216, 97.5% CI 2-sided [9.429 to 24.554]
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.548, 97.5% CI 2-sided [1.683 to 3.859]
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.055, 97.5% CI 2-sided [8.716 to 22.664]
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.536, 97.5% CI 2-sided [1.685 to 3.816]
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.106, 97.5% CI 2-sided [6.434 to 15.874]

11. Secondary Outcome: Percentage of Responders for Each Month, Except Month 3, in NMPP
Description: as for outcome 2
Time Frame: Months 1, 2, 4, 5, 6 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
percentage of participants
  Month 1 | 23.5 | 27.6 | 29.3
  Month 2 | 32.1 | 39.8 | 50.7
  Month 4 | 38.7 | 51.4 | 63.2
  Month 5 | 39.8 | 50.5 | 63.2
  Month 6 | 40.6 | 51.6 | 62.2
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.376, Regression, Logistic; Odds Ratio (OR) = 1.191, 97.5% CI 2-sided [0.765 to 1.855]
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.101, Regression, Logistic; Odds Ratio (OR) = 1.376, 97.5% CI 2-sided [0.890 to 2.127]
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.088, Regression, Logistic; Odds Ratio (OR) = 1.358, 97.5% CI 2-sided [0.909 to 2.029]
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.208, 97.5% CI 2-sided [1.488 to 3.278]
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.678, 97.5% CI 2-sided [1.136 to 2.477]
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.722, 97.5% CI 2-sided [1.832 to 4.044]
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.013, Regression, Logistic; Odds Ratio (OR) = 1.537, 97.5% CI 2-sided [1.042 to 2.267]
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.598, 97.5% CI 2-sided [1.750 to 3.857]
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.01, Regression, Logistic; Odds Ratio (OR) = 1.565, 97.5% CI 2-sided [1.062 to 2.306]
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.412, 97.5% CI 2-sided [1.630 to 3.570]

12. Secondary Outcome: Percentage of Responders at Each Month for DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe) as recorded in a daily electronic diary. The criteria for defining a participant as a responder included a reduction of -0.29 or greater from Baseline in DYSP as well as no increased rescue analgesic use for endometriosis-associated pain.
Time Frame: Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 262 | 168 | 171
percentage of participants
  Month 1: number analyzed (Participants) | 261 | 160 | 171
  Month 1 | 33.3 | 33.8 | 35.1
  Month 2 | 33.2 | 39.9 | 47.4
  Month 3: number analyzed (Participants) | 256 | 159 | 162
  Month 3 | 39.5 | 44.0 | 53.7
  Month 4: number analyzed (Participants) | 257 | 160 | 164
  Month 4 | 38.5 | 41.3 | 59.8
  Month 5: number analyzed (Participants) | 254 | 159 | 155
  Month 5 | 37.4 | 42.8 | 58.1
  Month 6: number analyzed (Participants) | 254 | 163 | 165
  Month 6 | 39.4 | 39.9 | 55.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.901, Regression, Logistic; Odds Ratio (OR) = 1.028, 97.5% CI 2-sided [0.624 to 1.693]
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.65, Regression, Logistic; Odds Ratio (OR) = 1.103, 97.5% CI 2-sided [0.680 to 1.789]
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.154, Regression, Logistic; Odds Ratio (OR) = 1.351, 97.5% CI 2-sided [0.841 to 2.170]
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.871, 97.5% CI 2-sided [1.175 to 2.979]
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.294, Regression, Logistic; Odds Ratio (OR) = 1.250, 97.5% CI 2-sided [0.776 to 2.013]
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.865, 97.5% CI 2-sided [1.163 to 2.989]
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.521, Regression, Logistic; Odds Ratio (OR) = 1.145, 97.5% CI 2-sided [0.713 to 1.839]
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.474, 97.5% CI 2-sided [1.544 to 3.963]
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.27, Regression, Logistic; Odds Ratio (OR) = 1.262, 97.5% CI 2-sided [0.787 to 2.023]
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.416, 97.5% CI 2-sided [1.500 to 3.891]
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.953, Regression, Logistic; Odds Ratio (OR) = 1.013, 97.5% CI 2-sided [0.631 to 1.624]
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.997, 97.5% CI 2-sided [1.253 to 3.183]

13. Secondary Outcome: Change From Baseline to Each Month, Except Month 6, in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline (Prior to administering study drug), Months 1, 2, 3, 4, 5 of Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
units on a scale
  Month 1 | -0.33 (0.044) | -0.86 (0.056) | -1.11 (0.056)
  Month 2: number analyzed (Participants) | 337 | 213 | 212
  Month 2 | -0.39 (0.042) | -0.84 (0.053) | -1.67 (0.053)
  Month 3: number analyzed (Participants) | 312 | 204 | 209
  Month 3 | -0.45 (0.042) | -0.97 (0.053) | -1.70 (0.052)
  Month 4: number analyzed (Participants) | 294 | 198 | 198
  Month 4 | -0.47 (0.044) | -1.05 (0.054) | -1.74 (0.054)
  Month 5: number analyzed (Participants) | 281 | 189 | 193
  Month 5 | -0.50 (0.045) | -0.99 (0.055) | -1.76 (0.055)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.53, 97.5% CI 2-sided [-0.69 to -0.37], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.78, 97.5% CI 2-sided [-0.94 to -0.62], Standard Error of Mean 0.071
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.44, 97.5% CI 2-sided [-0.6 to -0.29], Standard Error of Mean 0.068
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.27, 97.5% CI 2-sided [-1.43 to -1.12], Standard Error of Mean 0.068
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.53, 97.5% CI 2-sided [-0.68 to -0.37], Standard Error of Mean 0.068
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.25, 97.5% CI 2-sided [-1.4 to -1.09], Standard Error of Mean 0.067
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.58, 97.5% CI 2-sided [-0.73 to -0.42], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.27, 97.5% CI 2-sided [-1.42 to -1.11], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.49, 97.5% CI 2-sided [-0.65 to -0.33], Standard Error of Mean 0.071
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.26, 97.5% CI 2-sided [-1.42 to -1.10], Standard Error of Mean 0.071

14. Secondary Outcome: Percent Change From Baseline to Each Month in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 224
percentage change
  Month 1 | -14.36 (2.268) | -39.67 (2.886) | -53.68 (2.867)
  Month 2: number analyzed (Participants) | 337 | 213 | 211
  Month 2 | -17.36 (2.087) | -39.26 (2.629) | -80.68 (2.638)
  Month 3: number analyzed (Participants) | 312 | 204 | 208
  Month 3 | -20.58 (2.031) | -45.73 (2.528) | -82.52 (2.513)
  Month 4: number analyzed (Participants) | 294 | 198 | 198
  Month 4 | -21.55 (2.104) | -48.52 (2.601) | -83.92 (2.599)
  Month 5: number analyzed (Participants) | 281 | 189 | 193
  Month 5 | -22.63 (2.159) | -45.99 (2.664) | -85.53 (2.650)
  Month 6: number analyzed (Participants) | 273 | 185 | 187
  Month 6 | -23.81 (2.225) | -49.70 (2.738) | -80.43 (2.727)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -25.31, 97.5% CI 2-sided [-33.55 to -17.07], Standard Error of Mean 3.669
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -39.32, 97.5% CI 2-sided [-47.53 to -31.11], Standard Error of Mean 3.657
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -21.9, 97.5% CI 2-sided [-29.44 to -14.36], Standard Error of Mean 3.355
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -63.31, 97.5% CI 2-sided [-70.87 to -55.76], Standard Error of Mean 3.365
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -25.15, 97.5% CI 2-sided [-32.43 to -17.88], Standard Error of Mean 3.241
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -61.94, 97.5% CI 2-sided [-69.20 to -54.68], Standard Error of Mean 3.233
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -26.97, 97.5% CI 2-sided [-34.48 to -19.46], Standard Error of Mean 3.344
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -62.37, 97.5% CI 2-sided [-69.89 to -54.86], Standard Error of Mean 3.346
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -23.36, 97.5% CI 2-sided [-31.06 to -15.66], Standard Error of Mean 3.428
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -62.9, 97.5% CI 2-sided [-70.58 to -55.22], Standard Error of Mean 3.42
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -25.89, 97.5% CI 2-sided [-33.81 to -17.97], Standard Error of Mean 3.528
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -56.62, 97.5% CI 2-sided [-64.53 to -48.70], Standard Error of Mean 3.522

15. Secondary Outcome: Change From Baseline to Each Month, Except Month 6, in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Months 1, 2, 3, 4, 5 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
units on a scale
  Month 1 | -0.22 (0.025) | -0.24 (0.031) | -0.31 (0.031)
  Month 2: number analyzed (Participants) | 337 | 213 | 212
  Month 2 | -0.34 (0.027) | -0.41 (0.034) | -0.54 (0.034)
  Month 3: number analyzed (Participants) | 312 | 204 | 209
  Month 3 | -0.39 (0.031) | -0.50 (0.039) | -0.69 (0.039)
  Month 4: number analyzed (Participants) | 294 | 198 | 198
  Month 4 | -0.45 (0.033) | -0.54 (0.041) | -0.78 (0.041)
  Month 5: number analyzed (Participants) | 281 | 189 | 193
  Month 5 | -0.48 (0.034) | -0.58 (0.042) | -0.81 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.549, mixed-effects model; LS Mean of Difference = -0.02, 97.5% CI 2-sided [-0.11 to 0.07], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.02, mixed-effects model; LS Mean of Difference = -0.09, 97.5% CI 2-sided [-0.18 to 0.00], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.11, mixed-effects model; LS Mean of Difference = -0.07, 97.5% CI 2-sided [-0.17 to 0.03], Standard Error of Mean 0.044
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.20, 97.5% CI 2-sided [-0.30 to -0.11], Standard Error of Mean 0.043
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.041, mixed-effects model; LS Mean of Difference = -0.10, 97.5% CI 2-sided [-0.22 to 0.01], Standard Error of Mean 0.05
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.29, 97.5% CI 2-sided [-0.41 to -0.18], Standard Error of Mean 0.05
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.081, mixed-effects model; LS Mean of Difference = -0.09, 97.5% CI 2-sided [-0.21 to 0.03], Standard Error of Mean 0.052
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.33, 97.5% CI 2-sided [-0.45 to -0.22], Standard Error of Mean 0.052
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.062, mixed-effects model; LS Mean of Difference = -0.10, 97.5% CI 2-sided [-0.22 to 0.02], Standard Error of Mean 0.054
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.34, 97.5% CI 2-sided [-0.46 to -0.22], Standard Error of Mean 0.054

16. Secondary Outcome: Percent Change From Baseline to Each Month in the Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
percentage change
  Month 1 | -12.43 (1.814) | -15.47 (2.313) | -18.86 (2.288)
  Month 2: number analyzed (Participants) | 337 | 213 | 212
  Month 2 | -21.13 (1.836) | -26.30 (2.326) | -34.32 (2.316)
  Month 3: number analyzed (Participants) | 312 | 204 | 209
  Month 3 | -25.78 (2.104) | -32.63 (2.643) | -44.83 (2.625)
  Month 4: number analyzed (Participants) | 294 | 198 | 198
  Month 4 | -29.94 (2.170) | -36.19 (2.711) | -51.52 (2.696)
  Month 5: number analyzed (Participants) | 281 | 189 | 193
  Month 5 | -31.96 (2.214) | -38.17 (2.756) | -53.61 (2.737)
  Month 6: number analyzed (Participants) | 273 | 185 | 187
  Month 6 | -31.25 (2.349) | -42.09 (2.914) | -52.42 (2.897)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.301, mixed-effects model; LS Mean of Difference = -3.04, 97.5% CI 2-sided [-9.64 to 3.56], Standard Error of Mean 2.94
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.028, mixed-effects model; LS Mean of Difference = -6.43, 97.5% CI 2-sided [-12.99 to 0.13], Standard Error of Mean 2.92
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.082, mixed-effects model; LS Mean of Difference = -5.17, 97.5% CI 2-sided [-11.82 to 1.49], Standard Error of Mean 2.964
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -13.19, 97.5% CI 2-sided [-19.83 to -6.55], Standard Error of Mean 2.956
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.043, mixed-effects model; LS Mean of Difference = -6.84, 97.5% CI 2-sided [-14.43 to 0.75], Standard Error of Mean 3.379
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -19.05, 97.5% CI 2-sided [-26.61 to -11.49], Standard Error of Mean 3.364
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.072, mixed-effects model; LS Mean of Difference = -6.25, 97.5% CI 2-sided [-14.05 to 1.55], Standard Error of Mean 3.473
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -21.58, 97.5% CI 2-sided [-29.35 to -13.81], Standard Error of Mean 3.46
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.08, mixed-effects model; LS Mean of Difference = -6.21, 97.5% CI 2-sided [-14.15 to 1.73], Standard Error of Mean 3.536
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -21.66, 97.5% CI 2-sided [-29.56 to -13.75], Standard Error of Mean 3.52
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.004, mixed-effects model; LS Mean of Difference = -10.83, 97.5% CI 2-sided [-19.24 to -2.43], Standard Error of Mean 3.744
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -21.16, 97.5% CI 2-sided [-29.54 to -12.79], Standard Error of Mean 3.729

17. Secondary Outcome: Change From Baseline to Each Month, Except Month 3, in the Mean Pain Score of DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe).
Time Frame: Baseline, Months 1, 2, 4, 5, 6 of Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases. Participants who responded "not applicable" for the entire time point and at Baseline are excluded from the analysis. Participants with an assessment at given timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 261 | 161 | 171
units on a scale
  Month 1: number analyzed (Participants) | 261 | 160 | 171
  Month 1 | -0.21 (0.037) | -0.19 (0.046) | -0.26 (0.045)
  Month 2: number analyzed (Participants) | 247 | 161 | 162
  Month 2 | -0.25 (0.038) | -0.32 (0.047) | -0.49 (0.047)
  Month 4: number analyzed (Participants) | 212 | 143 | 146
  Month 4 | -0.35 (0.045) | -0.40 (0.055) | -0.63 (0.055)
  Month 5: number analyzed (Participants) | 196 | 137 | 133
  Month 5 | -0.39 (0.046) | -0.41 (0.056) | -0.70 (0.056)
  Month 6: number analyzed (Participants) | 189 | 137 | 137
  Month 6 | -0.36 (0.049) | -0.42 (0.058) | -0.69 (0.058)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.688, mixed-effects model; LS Mean of Difference = 0.02, 97.5% CI 2-sided [-0.11 to 0.16], Standard Error of Mean 0.059
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.431, mixed-effects model; LS Mean of Difference = -0.05, 97.5% CI 2-sided [-0.18 to 0.08], Standard Error of Mean 0.058
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.277, mixed-effects model; LS Mean of Difference = -0.07, 97.5% CI 2-sided [-0.20 to 0.07], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.24, 97.5% CI 2-sided [-0.37 to -0.10], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.494, mixed-effects model; LS Mean of Difference = -0.05, 97.5% CI 2-sided [-0.21 to 0.11], Standard Error of Mean 0.071
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.27, 97.5% CI 2-sided [-0.43 to -0.11], Standard Error of Mean 0.071
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.765, mixed-effects model; LS Mean of Difference = -0.02, 97.5% CI 2-sided [-0.18 to 0.14], Standard Error of Mean 0.072
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.31, 97.5% CI 2-sided [-0.47 to -0.15], Standard Error of Mean 0.073
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.468, mixed-effects model; LS Mean of Difference = -0.06, 97.5% CI 2-sided [-0.23 to 0.12], Standard Deviation 0.076
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.33, 97.5% CI 2-sided [-0.50 to -0.16], Standard Error of Mean 0.076

18. Secondary Outcome: Change From Baseline to Each Month, Except Months 3 and 6, in Analgesic Use Across Both Classes of Rescue Analgesics
Description: as for outcome 6
Time Frame: Baseline, Months 1, 2, 4, 5
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: number of pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
number of pills
  Month 1 | -0.20 (0.024) | -0.29 (0.031) | -0.32 (0.031)
  Month 2: number analyzed (Participants) | 337 | 213 | 212
  Month 2 | -0.25 (0.026) | -0.32 (0.033) | -0.44 (0.033)
  Month 4: number analyzed (Participants) | 294 | 198 | 198
  Month 4 | -0.29 (0.028) | -0.38 (0.035) | -0.51 (0.035)
  Month 5: number analyzed (Participants) | 281 | 189 | 193
  Month 5 | -0.32 (0.030) | -0.37 (0.038) | -0.54 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.029, mixed-effects model; LS Mean of Difference = -0.09, 97.5% CI 2-sided [-0.18 to 0.00], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.004, mixed-effects model; LS Mean of Difference = -0.11, 97.5% CI 2-sided [-0.20 to -0.03], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.076, mixed-effects model; LS Mean of Difference = -0.08, 97.5% CI 2-sided [-0.17 to 0.02], Standard Error of Mean 0.042
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.19, 97.5% CI 2-sided [-0.28 to -0.09], Standard Error of Mean 0.042
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.058, mixed-effects model; LS Mean of Difference = -0.09, 97.5% CI 2-sided [-0.19 to 0.02], Standard Error of Mean 0.045
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.22, 97.5% CI 2-sided [-0.32 to -0.12], Standard Error of Mean 0.045
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.284, mixed-effects model; LS Mean of Difference = -0.05, 97.5% CI 2-sided [-0.16 to 0.06], Standard Error of Mean 0.049
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.22, 97.5% CI 2-sided [-0.33 to -0.11], Standard Error of Mean 0.048

19. Secondary Outcome: Patient Global Impression of Change (PGIC) Questionnaire
Description: The PGIC questionnaire is a self-reported 7-point scale rating a participant's overall impression of change from 1 = very much improved to 7 = very much worse. Participants evaluated the change in their endometriosis-associated pain since initiation of study drug.
Time Frame: Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 337 | 214 | 215
units on a scale
  Month 1 | 3.49 (0.062) | 3.12 (0.078) | 2.84 (0.077)
  Month 2: number analyzed (Participants) | 331 | 210 | 210
  Month 2 | 3.24 (0.063) | 2.62 (0.079) | 2.15 (0.079)
  Month 3: number analyzed (Participants) | 332 | 211 | 209
  Month 3 | 3.16 (0.066) | 2.53 (0.083) | 2.02 (0.083)
  Month 4: number analyzed (Participants) | 329 | 212 | 212
  Month 4 | 3.19 (0.068) | 2.56 (0.085) | 1.97 (0.085)
  Month 5: number analyzed (Participants) | 333 | 212 | 213
  Month 5 | 3.23 (0.070) | 2.43 (0.088) | 1.98 (0.088)
  Month 6: number analyzed (Participants) | 325 | 213 | 210
  Month 6 | 3.22 (0.073) | 2.50 (0.090) | 1.95 (0.091)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.37, 95% CI 2-sided [-0.56 to -0.18], Standard Error of Mean 0.099
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.65, 95% CI 2-sided [-0.84 to -0.46], Standard Error of Mean 0.099
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.62, 95% CI 2-sided [-0.82 to -0.42], Standard Error of Mean 0.102
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.09, 95% CI 2-sided [-1.29 to -0.89], Standard Error of Mean 0.102
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.63, 95% CI 2-sided [-0.84 to -0.42], Standard Error of Mean 0.106
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.14, 95% CI 2-sided [-1.35 to -0.93], Standard Error of Mean 0.106
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.62, 95% CI 2-sided [-0.84 to -0.41], Standard Error of Mean 0.109
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.21, 95% CI 2-sided [-1.43 to -1.00], Standard Error of Mean 0.109
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.79, 95% CI 2-sided [-1.01 to -0.57], Standard Error of Mean 0.113
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.24, 95% CI 2-sided [-1.47 to -1.02], Standard Error of Mean 0.113
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.72, 95% CI 2-sided [-0.95 to -0.49], Standard Error of Mean 0.116
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.27, 95% CI 2-sided [-1.50 to -1.04], Standard Error of Mean 0.117

20. Secondary Outcome: Change From Baseline to Each Month, Except Month 3, in NRS Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Months 1, 2, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 358 | 221 | 225
units on a scale
  Month 1 | -0.78 (0.074) | -1.06 (0.094) | -1.23 (0.093)
  Month 2: number analyzed (Participants) | 336 | 213 | 212
  Month 2 | -1.08 (0.085) | -1.62 (0.108) | -2.04 (0.107)
  Month 4: number analyzed (Participants) | 294 | 198 | 198
  Month 4 | -1.49 (0.102) | -2.06 (0.128) | -2.84 (0.128)
  Month 5: number analyzed (Participants) | 281 | 189 | 193
  Month 5 | -1.58 (0.105) | -2.19 (0.131) | -2.95 (0.131)
  Month 6: number analyzed (Participants) | 273 | 185 | 187
  Month 6 | -1.60 (0.110) | -2.28 (0.137) | -2.87 (0.136)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.02, mixed-effects model; LS Mean of Difference = -0.28, 97.5% CI 2-sided [-0.55 to -0.01], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.45, 97.5% CI 2-sided [-0.72 to -0.18], Standard Error of Mean 0.119
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.54, 97.5% CI 2-sided [-0.85 to -0.23], Standard Error of Mean 0.137
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.96, 97.5% CI 2-sided [-1.27 to -0.65], Standard Error of Mean 0.137
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.58, 97.5% CI 2-sided [-0.95 to -0.21], Standard Error of Mean 0.164
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.36, 97.5% CI 2-sided [-1.72 to -0.99], Standard Error of Mean 0.164
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.61, 97.5% CI 2-sided [-0.99 to -0.23], Standard Error of Mean 0.168
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.37, 97.5% CI 2-sided [-1.75 to -1.00], Standard Error of Mean 0.168
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.69, 97.5% CI 2-sided [-1.08 to -0.30], Standard Error of Mean 0.175
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.28, 97.5% CI 2-sided [-1.67 to -0.89], Standard Error of Mean 0.175

21. Secondary Outcome: Change From Baseline to Each Scheduled Assessment in the Pain Domain of Endometriosis Health Profile-30 (EHP-30) Questionnaire Scores
Description: The EHP-30 is a disease-specific self-administered questionnaire used to measure health-related quality of life in women with endometriosis. Each domain is calculated on a scale from 0 = best possible health status to 100 = worst possible health status.
Time Frame: Baseline, Months 1, 3, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 331 | 213 | 213
units on a scale
  Month 1 | -15.20 (0.971) | -19.40 (1.210) | -22.75 (1.211)
  Month 3: number analyzed (Participants) | 304 | 203 | 200
  Month 3 | -19.29 (1.103) | -26.62 (1.349) | -34.72 (1.360)
  Month 6: number analyzed (Participants) | 230 | 161 | 167
  Month 6 | -19.53 (1.340) | -28.23 (1.601) | -36.44 (1.572)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.007, ANCOVA; Difference in LS Means = -4.2, 95% CI 2-sided [-7.25 to -1.16], Standard Error of Mean 1.55
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -7.55, 95% CI 2-sided [-10.6 to -4.50], Standard Error of Mean 1.55
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -7.33, 95% CI 2-sided [-10.75 to -3.91], Standard Error of Mean 1.74
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -15.43, 95% CI 2-sided [-18.87 to -11.99], Standard Error of Mean 1.75
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -8.7, 95% CI 2-sided [-12.81 to -4.60], Standard Error of Mean 2.09
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -16.92, 95% CI 2-sided [-20.98 to -12.86], Standard Error of Mean 2.07

22. Secondary Outcome: Change From Baseline to Each Scheduled Assessment in the Sexual Intercourse Domain of EHP-30 Questionnaire Scores
Description: as for outcome 21
Time Frame: Baseline, Months 1, 3, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 226 | 150 | 155
units on a scale
  Month 1 | -9.89 (1.229) | -10.46 (1.510) | -14.29 (1.484)
  Month 3: number analyzed (Participants) | 221 | 139 | 146
  Month 3 | -14.51 (1.502) | -17.26 (1.895) | -25.20 (1.848)
  Month 6: number analyzed (Participants) | 152 | 111 | 124
  Month 6 | -14.14 (1.891) | -17.07 (2.215) | -28.24 (2.095)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.77, ANCOVA; Difference in LS Means = -0.57, 95% CI 2-sided [-4.40 to 3.26], Standard Error of Mean 1.95
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.023, ANCOVA; Difference in LS Means = -4.40, 95% CI 2-sided [-8.19 to -0.61], Standard Error of Mean 1.93
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.257, ANCOVA; Difference in LS Means = -2.74, 95% CI 2-sided [-7.50 to 2.01], Standard Error of Mean 2.42
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -10.69, 95% CI 2-sided [-15.37 to -6.01], Standard Error of Mean 2.38
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.315, ANCOVA; Difference in LS Means = -2.93, 95% CI 2-sided [-8.66 to 2.80], Standard Error of Mean 2.91
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -14.1, 95% CI 2-sided [-19.64 to -8.55], Standard Error of Mean 2.82

23. Secondary Outcome: Change From Baseline to Each Month in Health Related Productivity Questionnaire (HRPQ): Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the workplace due to absenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 239 | 150 | 146
hours
  Month 1 | -0.61 (0.267) | -1.62 (0.336) | -1.56 (0.341)
  Month 2: number analyzed (Participants) | 229 | 142 | 142
  Month 2 | -0.82 (0.246) | -1.80 (0.312) | -2.25 (0.312)
  Month 3: number analyzed (Participants) | 217 | 137 | 138
  Month 3 | -0.76 (0.268) | -1.43 (0.338) | -2.17 (0.336)
  Month 4: number analyzed (Participants) | 198 | 133 | 138
  Month 4 | -0.55 (0.355) | -1.81 (0.434) | -2.03 (0.426)
  Month 5: number analyzed (Participants) | 190 | 132 | 132
  Month 5 | -0.85 (0.209) | -1.58 (0.251) | -1.96 (0.251)
  Month 6: number analyzed (Participants) | 142 | 93 | 98
  Month 6 | -0.76 (0.246) | -1.34 (0.303) | -1.67 (0.296)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.019, ANCOVA; Difference in LS Means = -1.01, 95% CI 2-sided [-1.86 to -0.17], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.028, ANCOVA; Difference in LS Means = -0.95, 95% CI 2-sided [-1.80 to -0.10], Standard Error of Mean 0.433
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.014, ANCOVA; Difference in LS Means = -0.98, 95% CI 2-sided [-1.76 to -0.20], Standard Error of Mean 0.397
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.44, 95% CI 2-sided [-2.22 to -0.65], Standard Error of Mean 0.397
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.121, ANCOVA; Difference in LS Means = -0.67, 95% CI 2-sided [-1.52 to 0.18], Standard Error of Mean 0.432
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p = 0.001, ANCOVA; Difference in LS Means = -1.41, 95% CI 2-sided [-2.25 to -0.56], Standard Error of Mean 0.431
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.026, ANCOVA; Difference in LS Means = -1.25, 95% CI 2-sided [-2.35 to -0.15], Standard Error of Mean 0.561
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p = 0.008, ANCOVA; Difference in LS Means = -1.48, 95% CI 2-sided [-2.57 to -0.39], Standard Error of Mean 0.555
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.027, ANCOVA; Difference in LS Means = -0.73, 95% CI 2-sided [-1.37 to -0.08], Standard Error of Mean 0.327
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.11, 95% CI 2-sided [-1.75 to -0.47], Standard Error of Mean 0.327
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.143, ANCOVA; Difference in LS Means = -0.57, 95% CI 2-sided [-1.34 to 0.20], Standard Error of Mean 0.391
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p = 0.019, ANCOVA; Difference in LS Means = -0.91, 95% CI 2-sided [-1.67 to -0.15], Standard Error of Mean 0.385

24. Secondary Outcome: Change From Baseline to Each Month in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the household due to absenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 272 | 178 | 187
hours
  Month 1 | -1.45 (0.261) | -2.08 (0.322) | -2.30 (0.315)
  Month 2: number analyzed (Participants) | 253 | 172 | 169
  Month 2 | -1.63 (0.269) | -2.75 (0.327) | -3.06 (0.330)
  Month 3: number analyzed (Participants) | 248 | 164 | 167
  Month 3 | -2.03 (0.274) | -2.95 (0.336) | -2.94 (0.333)
  Month 4: number analyzed (Participants) | 219 | 143 | 169
  Month 4 | -2.21 (0.285) | -2.55 (0.353) | -3.54 (0.324)
  Month 5: number analyzed (Participants) | 216 | 151 | 156
  Month 5 | -1.87 (0.284) | -2.99 (0.340) | -3.51 (0.334)
  Month 6: number analyzed (Participants) | 158 | 109 | 131
  Month 6 | -1.89 (0.306) | -2.61 (0.368) | -3.34 (0.336)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.131, ANCOVA; Difference in LS Means = -0.63, 95% CI 2-sided [-1.44 to 0.19], Standard Error of Mean 0.415
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.037, ANCOVA; Difference in LS Means = -0.85, 95% CI 2-sided [-1.65 to -0.05], Standard Error of Mean 0.409
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.008, ANCOVA; Difference in LS Means = -1.12, 95% CI 2-sided [-1.96 to -0.29], Standard Error of Mean 0.423
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.44, 95% CI 2-sided [-2.27 to -0.60], Standard Error of Mean 0.426
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.036, ANCOVA; Difference in LS Means = -0.91, 95% CI 2-sided [-1.76 to -0.06], Standard Error of Mean 0.434
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p = 0.035, ANCOVA; Difference in LS Means = -0.91, 95% CI 2-sided [-1.76 to -0.06], Standard Error of Mean 0.431
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.452, ANCOVA; Difference in LS Means = -0.34, 95% CI 2-sided [-1.23 to 0.55], Standard Error of Mean 0.453
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -1.33, 95% CI 2-sided [-2.18 to -0.48], Standard Error of Mean 0.432
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.012, ANCOVA; Difference in LS Means = -1.12, 95% CI 2-sided [-1.99 to -0.25], Standard Error of Mean 0.443
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.64, 95% CI 2-sided [-2.5 to -0.78], Standard Error of Mean 0.439
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.13, ANCOVA; Difference in LS Means = -0.73, 95% CI 2-sided [-1.67 to 0.21], Standard Error of Mean 0.478
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p = 0.001, ANCOVA; Difference in LS Means = -1.45, 95% CI 2-sided [-2.34 to -0.56], Standard Error of Mean 0.454

25. Secondary Outcome: Change From Baseline to Each Month in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the workplace due to presenteeism [working while sick]) in the 7 days prior to survey administration.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 235 | 145 | 143
hours
  Month 1 | -1.60 (0.623) | -2.94 (0.793) | -4.69 (0.798)
  Month 2: number analyzed (Participants) | 223 | 138 | 137
  Month 2 | -3.43 (0.621) | -4.74 (0.790) | -7.08 (0.792)
  Month 3: number analyzed (Participants) | 213 | 134 | 133
  Month 3 | -4.07 (0.633) | -6.10 (0.799) | -7.27 (0.801)
  Month 4: number analyzed (Participants) | 195 | 129 | 132
  Month 4 | -4.58 (0.629) | -6.21 (0.774) | -9.35 (0.764)
  Month 5: number analyzed (Participants) | 186 | 127 | 125
  Month 5 | -4.37 (0.618) | -6.66 (0.747) | -9.51 (0.753)
  Month 6: number analyzed (Participants) | 142 | 90 | 95
  Month 6 | -6.11 (0.692) | -7.08 (0.869) | -9.13 (0.845)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.186, ANCOVA; Difference in LS Means = -1.34, 95% CI 2-sided [-3.32 to 0.65], Standard Error of Mean 1.01
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -3.09, 95% CI 2-sided [-5.08 to -1.10], Standard Error of Mean 1.013
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.195, ANCOVA; Difference in LS Means = -1.31, 95% CI 2-sided [-3.28 to 0.67], Standard Error of Mean 1.005
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.65, 95% CI 2-sided [-5.63 to -1.67], Standard Error of Mean 1.007
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.047, ANCOVA; Difference in LS Means = -2.03, 95% CI 2-sided [-4.03 to -0.02], Standard Error of Mean 1.02
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -3.2, 95% CI 2-sided [-5.21 to -1.19], Standard Error of Mean 1.021
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.103, ANCOVA; Difference in LS Means = -1.63, 95% CI 2-sided [-3.59 to 0.33], Standard Error of Mean 0.998
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -4.78, 95% CI 2-sided [-6.72 to -2.83], Standard Error of Mean 0.99
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.019, ANCOVA; Difference in LS Means = -2.29, 95% CI 2-sided [-4.20 to -0.38], Standard Error of Mean 0.970
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -5.14, 95% CI 2-sided [-7.06 to -3.22], Standard Error of Mean 0.975
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.383, ANCOVA; Difference in LS Means = -0.97, 95% CI 2-sided [-3.16 to 1.22], Standard Error of Mean 1.112
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p = 0.006, ANCOVA; Difference in LS Means = -3.02, 95% CI 2-sided [-5.17 to -0.87], Standard Error of Mean 1.092

26. Secondary Outcome: Change From Baseline to Each Month in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the household due to presenteeism [working while sick]) in the 7 days prior to survey administration.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 266 | 175 | 185
hours
  Month 1 | -0.71 (0.266) | -0.69 (0.327) | -0.72 (0.319)
  Month 2: number analyzed (Participants) | 249 | 168 | 163
  Month 2 | -1.06 (0.247) | -1.28 (0.301) | -1.46 (0.305)
  Month 3: number analyzed (Participants) | 246 | 162 | 162
  Month 3 | -1.31 (0.318) | -0.88 (0.392) | -1.46 (0.392)
  Month 4: number analyzed (Participants) | 218 | 141 | 166
  Month 4 | -1.26 (0.308) | -1.19 (0.383) | -2.19 (0.353)
  Month 5: number analyzed (Participants) | 214 | 148 | 152
  Month 5 | -0.78 (0.406) | -1.68 (0.488) | -1.69 (0.482)
  Month 6: number analyzed (Participants) | 156 | 108 | 128
  Month 6 | -1.44 (0.318) | -2.27 (0.383) | -2.29 (0.351)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.975, ANCOVA; Difference in LS Means = 0.01, 95% CI 2-sided [-0.81 to 0.84], Standard Error of Mean 0.422
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.969, ANCOVA; Difference in LS Means = -0.02, 95% CI 2-sided [-0.83 to 0.80], Standard Error of Mean 0.415
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.569, ANCOVA; Difference in LS Means = -0.22, 95% CI 2-sided [-0.99 to 0.54], Standard Error of Mean 0.389
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p = 0.311, ANCOVA; Difference in LS Means = -0.4, 95% CI 2-sided [-1.17 to 0.37], Standard Error of Mean 0.393
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.398, ANCOVA; Difference in LS Means = 0.43, 95% CI 2-sided [-0.56 to 1.42], Standard Error of Mean 0.505
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p = 0.761, ANCOVA; Difference in LS Means = -0.15, 95% CI 2-sided [-1.15 to 0.84], Standard Error of Mean 0.505
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.874, ANCOVA; Difference in LS Means = 0.08, 95% CI 2-sided [-0.89 to 1.04], Standard Error of Mean 0.491
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p = 0.048, ANCOVA; Difference in LS Means = -0.93, 95% CI 2-sided [-1.85 to -0.01], Standard Error of Mean 0.468
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.16, ANCOVA; Difference in LS Means = -0.89, 95% CI 2-sided [-2.14 to 0.35], Standard Error of Mean 0.635
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p = 0.152, ANCOVA; Difference in LS Means = -0.9, 95% CI 2-sided [-2.14 to 0.33], Standard Error of Mean 0.63
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.095, ANCOVA; Difference in LS Means = -0.83, 95% CI 2-sided [-1.81 to 0.15], Standard Error of Mean 0.498
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p = 0.071, ANCOVA; Difference in LS Means = -0.86, 95% CI 2-sided [-1.79 to 0.07], Standard Error of Mean 0.474

27. Secondary Outcome: Change From Baseline to Each Month in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the workplace due to absenteeism and presenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 239 | 150 | 146
hours
  Month 1 | -2.19 (0.686) | -4.02 (0.865) | -5.91 (0.875)
  Month 2: number analyzed (Participants) | 229 | 142 | 142
  Month 2 | -4.25 (0.674) | -6.27 (0.856) | -9.36 (0.854)
  Month 3: number analyzed (Participants) | 217 | 137 | 138
  Month 3 | -4.66 (0.708) | -7.31 (0.891) | -9.30 (0.886)
  Month 4: number analyzed (Participants) | 198 | 133 | 138
  Month 4 | -4.87 (0.721) | -7.58 (0.879) | -11.14 (0.862)
  Month 5: number analyzed (Participants) | 190 | 132 | 132
  Month 5 | -5.32 (0.701) | -7.81 (0.839) | -11.15 (0.839)
  Month 6: number analyzed (Participants) | 142 | 93 | 98
  Month 6 | -6.73 (0.793) | -8.01 (0.980) | -10.70 (0.953)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.098, ANCOVA; Difference in LS Means = -1.83, 95% CI 2-sided [-4.01 to 0.34], Standard Error of Mean 1.106
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.72, 95% CI 2-sided [-5.91 to -1.54], Standard Error of Mean 1.113
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.065, ANCOVA; Difference in LS Means = -2.02, 95% CI 2-sided [-4.16 to 0.13], Standard Error of Mean 1.091
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -5.1, 95% CI 2-sided [-7.24 to -2.96], Standard Error of Mean 1.089
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.02, ANCOVA; Difference in LS Means = -2.65, 95% CI 2-sided [-4.89 to -0.41], Standard Error of Mean 1.14
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -4.64, 95% CI 2-sided [-6.87 to -2.41], Standard Error of Mean 1.135
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.017, ANCOVA; Difference in LS Means = -2.72, 95% CI 2-sided [-4.95 to -0.48], Standard Error of Mean 1.138
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -6.27, 95% CI 2-sided [-8.48 to -4.06], Standard Error of Mean 1.124
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.023, ANCOVA; Difference in LS Means = -2.49, 95% CI 2-sided [-4.64 to -0.34], Standard Error of Mean 1.095
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -5.83, 95% CI 2-sided [-7.98 to -3.68], Standard Error of Mean 1.095
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.311, ANCOVA; Difference in LS Means = -1.28, 95% CI 2-sided [-3.77 to 1.20], Standard Error of Mean 1.264
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p = 0.001, ANCOVA; Difference in LS Means = -3.97, 95% CI 2-sided [-6.42 to -1.53], Standard Error of Mean 1.241

28. Secondary Outcome: Change From Baseline to Each Month in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the household due to absenteeism and presenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 272 | 178 | 187
hours
  Month 1 | -2.18 (0.390) | -2.78 (0.482) | -2.89 (0.470)
  Month 2: number analyzed (Participants) | 253 | 172 | 169
  Month 2 | -2.71 (0.415) | -4.04 (0.503) | -4.48 (0.508)
  Month 3: number analyzed (Participants) | 248 | 164 | 167
  Month 3 | -3.37 (0.448) | -3.84 (0.551) | -4.34 (0.546)
  Month 4: number analyzed (Participants) | 219 | 143 | 169
  Month 4 | -3.46 (0.463) | -3.77 (0.574) | -5.64 (0.528)
  Month 5: number analyzed (Participants) | 216 | 151 | 156
  Month 5 | -2.62 (0.549) | -4.67 (0.657) | -5.16 (0.646)
  Month 6: number analyzed (Participants) | 158 | 109 | 131
  Month 6 | -3.30 (0.497) | -4.89 (0.598) | -5.58 (0.546)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Month 1; Test type: Superiority; p = 0.335, ANCOVA; Difference in LS Means = -0.60, 95% CI 2-sided [-1.81 to 0.62], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Month 1; Test type: Superiority; p = 0.242, ANCOVA; Difference in LS Means = -0.72, 95% CI 2-sided [-1.91 to 0.48], Standard Error of Mean 0.611
Statistical Analysis 3: Comparison: Placebo vs Elagolix 150 mg QD; Month 2; Test type: Superiority; p = 0.042, ANCOVA; Difference in LS Means = -1.33, 95% CI 2-sided [-2.61 to -0.05], Standard Error of Mean 0.652
Statistical Analysis 4: Comparison: Placebo vs Elagolix 200 mg BID; Month 2; Test type: Superiority; p = 0.007, ANCOVA; Difference in LS Means = -1.77, 95% CI 2-sided [-3.06 to -0.48], Standard Error of Mean 0.656
Statistical Analysis 5: Comparison: Placebo vs Elagolix 150 mg QD; Month 3; Test type: Superiority; p = 0.503, ANCOVA; Difference in LS Means = -0.48, 95% CI 2-sided [-1.87 to 0.92], Standard Error of Mean 0.71
Statistical Analysis 6: Comparison: Placebo vs Elagolix 200 mg BID; Month 3; Test type: Superiority; p = 0.169, ANCOVA; Difference in LS Means = -0.97, 95% CI 2-sided [-2.36 to 0.41], Standard Error of Mean 0.707
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg QD; Month 4; Test type: Superiority; p = 0.675, ANCOVA; Difference in LS Means = -0.31, 95% CI 2-sided [-1.76 to 1.14], Standard Error of Mean 0.737
Statistical Analysis 8: Comparison: Placebo vs Elagolix 200 mg BID; Month 4; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -2.17, 95% CI 2-sided [-3.55 to -0.79], Standard Error of Mean 0.703
Statistical Analysis 9: Comparison: Placebo vs Elagolix 150 mg QD; Month 5; Test type: Superiority; p = 0.017, ANCOVA; Difference in LS Means = -2.04, 95% CI 2-sided [-3.72 to -0.36], Standard Error of Mean 0.856
Statistical Analysis 10: Comparison: Placebo vs Elagolix 200 mg BID; Month 5; Test type: Superiority; p = 0.003, ANCOVA; Difference in LS Means = -2.54, 95% CI 2-sided [-4.21 to -0.87], Standard Error of Mean 0.848
Statistical Analysis 11: Comparison: Placebo vs Elagolix 150 mg QD; Month 6; Test type: Superiority; p = 0.042, ANCOVA; Difference in LS Means = -1.59, 95% CI 2-sided [-3.12 to -0.06], Standard Error of Mean 0.778
Statistical Analysis 12: Comparison: Placebo vs Elagolix 200 mg BID; Month 6; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -2.28, 95% CI 2-sided [-3.73 to -0.83], Standard Error of Mean 0.738

29. Secondary Outcome: Number of Participants With Endometriosis-Related Non-Study Health Visits During the Treatment Period
Description: This is assessed using Health Resource Utilization Questionnaire (HRUQ).
Time Frame: Months 1, 2, 3, 4, 5, 6 of Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 360 | 226 | 229
Participants
  Baseline | 99 | 53 | 57
  Month 1 | 93 | 47 | 54
  Month 2 | 72 | 42 | 43
  Month 3 | 54 | 46 | 40
  Month 4 | 62 | 39 | 43
  Month 5 | 56 | 31 | 30
  Month 6 | 39 | 27 | 25
  Overall | 201 | 124 | 131

30. Secondary Outcome: Number of Days of Hospitalization
Description: This is assessed using HRUQ.
Time Frame: Up to Month 6 of Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Includes participants who were hospitalized during the Treatment Period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 18 | 16 | 12
days | 3.2 (2.18) | 3.3 (3.52) | 2.2 (1.27)

31. Secondary Outcome: Number of Participants With Emergency Room/Outpatient Procedures During the Treatment Period, by Type
Description: This is assessed using HRUQ.
Time Frame: Up to Month 6 of Treatment Period
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 360 | 226 | 229
Participants
  All Categories | 37 | 28 | 22
  Abdominal Hysterectomy | 0 | 0 | 0
  Angiography | 0 | 1 | 0
  Arthroscopy | 0 | 0 | 1
  Biopsy | 0 | 1 | 1
  Blood Draw | 12 | 13 | 4
  Colposcopy | 0 | 0 | 0
  Consultation | 1 | 5 | 1
  CT Scan | 7 | 10 | 5
  Diagnostic Laparoscopy | 0 | 0 | 0
  Electrocardiogram | 4 | 2 | 0
  Endometrial Ablation | 0 | 0 | 0
  Histological Exam | 0 | 0 | 0
  Intrauterine Insemination | 0 | 0 | 0
  In Vitro Fertilization | 0 | 0 | 0
  Laparoscopic Hysterectomy | 0 | 0 | 0
  Laparotomy | 0 | 0 | 0
  Magnetic Resonance Imaging | 0 | 2 | 0
  Oophorectomy | 0 | 0 | 0
  Pelvic Exam | 3 | 0 | 2
  Physical Examination | 18 | 16 | 14
  Surgery for Adhesions | 0 | 0 | 0
  Therapeutic Laparoscopy | 0 | 0 | 0
  Transfusion | 0 | 0 | 0
  Ultrasound | 9 | 3 | 2
  Urine Test | 8 | 7 | 6
  Vaginal Hysterectomy | 0 | 0 | 0
  X-Ray | 12 | 11 | 7
  Other (Not Specified) | 13 | 4 | 4

ADVERSE EVENTS:
Time Frame: From first dose of study treatment through 6 months of treatment plus up to 12 months of follow-up.
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
All-Cause Mortality (participants affected / at risk) | 0/360 | 1/226 | 0/229
Serious Adverse Events (participants affected / at risk) | 12/360 | 12/226 | 5/229
Other Adverse Events (participants affected / at risk) | 158/360 | 128/226 | 162/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=360) | Elagolix 150 mg QD (N=226) | Elagolix 200 mg BID (N=229)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
PHARYNGEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
JAW CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS COMPLETE (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
PERINEAL PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
BLOOD PRESSURE FLUCTUATION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=360) | Elagolix 150 mg QD (N=226) | Elagolix 200 mg BID (N=229)
DIARRHOEA (Gastrointestinal disorders) | 18 (18) | 8 (8) | 11 (11)
NAUSEA (Gastrointestinal disorders) | 40 (40) | 26 (26) | 36 (36)
NASOPHARYNGITIS (Infections and infestations) | 21 (21) | 15 (15) | 16 (16)
SINUSITIS (Infections and infestations) | 14 (14) | 10 (10) | 15 (15)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 (16) | 11 (11) | 12 (12)
URINARY TRACT INFECTION (Infections and infestations) | 26 (26) | 10 (10) | 19 (19)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7) | 16 (16)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 (15) | 8 (8) | 13 (13)
HEADACHE (Nervous system disorders) | 50 (50) | 42 (42) | 52 (52)
INSOMNIA (Psychiatric disorders) | 12 (12) | 13 (13) | 24 (24)
MOOD SWINGS (Psychiatric disorders) | 8 (8) | 13 (13) | 6 (6)
AMENORRHOEA (Reproductive system and breast disorders) | 1 (1) | 11 (11) | 20 (20)
HOT FLUSH (Vascular disorders) | 37 (37) | 51 (51) | 109 (109)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.